CLINICAL TRIAL: NCT05637255
Title: A Randomized, Double Masked, Parallel Group, Dose-finding Study to Evaluate SYL1801 in Patients With Neovascular AMD
Brief Title: A Randomized, Double Masked, Parallel Group, Dose-finding Study to Evaluate SYL1801 in Patients With Neovascular Age-related Macular Degeneration (AMD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYL1801_II; 2022-000214-34 (EudraCT Number)
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Wet Macular Degeneration; Neovascular Age-related Macular Degeneration; Macular Degeneration
Keywords: siRNA; oligonucleotide
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SYL1801 ophthalmic solution Low Dose once daily (Experimental): 42 treatment days
  Interventions: Drug: SYL1801
- SYL1801 ophthalmic solution Middle Dose once daily (Experimental): 42 treatment days
  Interventions: Drug: SYL1801
- SYL1801 ophthalmic solution High Dose once daily (Experimental): 42 treatment days
  Interventions: Drug: SYL1801

INTERVENTIONS:
Drug: SYL1801 — 1 drop in the eligible eye

SUMMARY:
The goal of this clinical trial is to compare the safety and effect on visual acuity of three different doses of SYL1801 eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Active subfoveal or juxtafoveal choroidal neovascularization secondary to AMD
* Best Corrected Visual Acuity (BCVA) between 70-25 letters (ETDRS) at Screening
* Intraretinal or subretinal fluid
* Central Subfield Thickness > 300 µm

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test.
* Females of childbearing potential who will not use a medically acceptable contraceptive method
* Current, previous chronic or recurrent condition according to the investigator's judgement.
* Concomitant treatment or prior ocular procedure or surgery, or alteration of the dose of systemic medications
* Concurrent disease in the study eye
* Previous treatment with systemic anti-Vascular Endothelial Growing Factor (Anti-VEGF) drugs or pro-VEGF treatments
* Concurrent disease in the study eye, other than AMD

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-07-22 (Estimated); Study Completion 2023-11-22 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on visual acuity on Day 42 after last instillation of the assigned dose level | 42 days after first administration
  ETDRS chart

SECONDARY OUTCOMES:
Proportion of subjects within each cohort who maintained visual acuity on Day 42 after last instillation of the assigned dose level | 42 days after first administration
  ETDRS chart
Proportion of subjects within each cohort who gained visual acuity on Day 42 after last instillation of the assigned dose level | Through study completion, up to 42 days
  ETDRS chart
Proportion of subjects within each cohort who needed rescue medication at any point of the study | Through study completion, up to 42 days
Change from Baseline on flow area on Day 42 after last instillation of the assigned | 42 days after first administration
  Optical Coherence Tomography Angiography (OCTA)
Change from Screening on leakage area on Day 42 after last instillation of the assigned | 43 days after first administration
  Fluorescein Angiography
Change from Baseline on intraocular pressure (IOP) | 42 days after first administration
  Tonometry
Adverse Event Evaluation | Through study completion, up to 42 days

CONTACTS AND LOCATIONS:
Locations (15):
- Czechia (7):
  - SYL1801 Investigative Site, Brno
  - SYL1801 Investigative Site, Chomutov
  - SYL1801 Investigative Site, Frýdek-Místek
  - SYL1801 Investigative Site, Kyjov
  - SYL1801 Investigative Site, Liberec
  - SYL1801 Investigative Site, Ostrava
  - SYL1801 Investigative Site, Prague
- Poland (4):
  - SYL1801 Investigative Site, Gdansk
  - SYL1801 Investigative Site, Krakow
  - SYL1801 Investigative Site, Rzeszów
  - SYL1801 Investigative Site, Warsaw
- Slovakia (4):
  - SYL1801 Investigative Site, Bratislava
  - SYL1801 Investigative Site, Košice
  - SYL1801 Investigative Site, Poprad
  - SYL1801 Investigative Site, Žilina